CLINICAL TRIAL: NCT04883346
Title: Phase II Trial of Liraglutide (Saxenda(R), Novo Nordisk) in Adolescents With Obesity After Sleeve Gastrectomy: A Pilot Open-Label Study
Brief Title: Liraglutide (Saxenda(R)) in Adolescents With Obesity After Sleeve Gastrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000241; 000241-CH (Other: NIH Clinical Center)
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-05-16

CONDITIONS: Obesity; Status Post Sleeve Gastrectomy
Keywords: Children; glucagon-like peptide; Weight Loss; pharmacotherapy for obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liraglutide (Experimental): Treated with Liraglutide
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide by subcutaneous injection administered daily. Dose will be initiated at 0.6mg per day and increased to a maximum of 3.0 mg per day as tolerated.
  Other Names: Saxenda

SUMMARY:
Background:

Metabolic Bariatric Surgery, including a surgery called vertical sleeve gastrectomy, is the most effective weight loss treatment for severe obesity. However, many adolescents who have this surgery still have obesity 1 year later or regain weight. Researchers want to see if a drug can help.

Objective:

To learn if liraglutide can help adolescents who still have obesity 1 year or more after vertical sleeve gastrectomy lose additional weight.

Eligibility:

Healthy adolescents ages 12-20.99 years who are 1-10 years post vertical sleeve gastrectomy and have a BMI of 30 kg/m2 or >=95th percentile for age and sex.

Design:

Participants will be screened with:

Medical history

Physical exam

Questionnaires about their mood and feelings about their weight

Blood and urine tests

Nutrition counseling. They will keep a diet log.

A test where they view and respond to pictures of food

Wrist accelerometer set-up. They will wear an accelerometer (a device like a watch) on their wrist for 14 days. It will measure their physical activity.

Some screening tests will be repeated during the study.

Participants will have an oral glucose tolerance test. They will ingest a sweet liquid. Blood samples will be taken.

Participants will take liraglutide daily for 16 weeks. They will learn how to inject it under their skin.

Participants will have a body scan to measure muscle and fat.

Participants will be invited to eat as much as they want at a buffet meal at NIH. How much food they eat will be calculated. They will assess their appetite and mood before and after the meal.

Participation will last for 7 months. Participants will have up to 7 study visits....

DETAILED DESCRIPTION:
Study Description:

This trial is an open-label Phase II non-randomized pilot study conducted at the NIH Clinical Center to investigate the efficacy of daily subcutaneous injection of liraglutide, a glucagon-like peptide-1 (GLP1) analogue to promote reduction of body mass index (BMI) in adolescents who continue to have obesity (BMI (Bullet)30 or BMI >=95th percentile for age and sex) 1 year or more after vertical sleeve gastrectomy (SG). We hypothesize that administration of liraglutide will be associated with reduction in BMI in such adolescents.

Objectives:

Primary objective: To determine the effect size for the change in BMI of liraglutide 3.0 mg daily subcutaneously at 16 weeks in adolescents who have obesity after SG, in order to use the observed changes to determine the sample size of a subsequent randomized, controlled investigation.

Hypothesis:

The Primary Endpoint is estimation of required sample size for a later randomized controlled trial through calculation of effect size for change in body mass index (BMI) from baseline to 16 weeks of liraglutide. The hypothesis is: The data will be sufficient to calculate the effect size for change in BMI from baseline to 16 weeks for a 2-group experiment (placebo versus liraglutide).

Secondary objectives:

To study the effects of 16 weeks of liraglutide 3.0 mg subcutaneously on change in mean BMI and fat mass in adolescents who underwent vertical sleeve gastrectomy (SG) >=1y prior to study initiation but still have obesity or have a recrudescence of obesity despite surgery. To compare the effects of liraglutide on BMI and fat mass in enrolled participants who had a poor initial response to SG (<20% BMI reduction at BMI nadir) vs. those with a typical post-SG weight loss (>=20% BMI reduction at BMI nadir).

Additional Objectives:

To examine the effects of daily subcutaneous liraglutide in enrolled participants on changes in body composition, metabolic syndrome markers, energy intake, glucose tolerance, gastrointestinal (GI)

hormone concentrations, appetite, free living physical activity, mood, suicidality, weight related quality of life, self-perception of body image, and secretome.

Endpoints:

Primary Endpoint: Estimation of required sample size for a later RCT through calculation of effect size for change in body mass index (BMI) from baseline to 16 weeks of liraglutide.

Key Secondary Endpoints:

Changes in BMI and fat mass after 16 weeks of liraglutide Comparison of changes in BMI and fat mass after 16 weeks of liraglutide in participants who had a poor initial response to SG (<20% BMI reduction at BMI nadir) vs. those with a typical post-S weight loss (>=20% BMI reduction at BMI nadir) Tolerability and safety of liraglutide 3.0 mg.

Additional (exploratory) Endpoints: Change from baseline to 16 weeks of liraglutide in:

1. Proportion reducing BMI by at least 5% and 10%
2. BMI standard deviation score for age and sex (BMIz)
3. Body weight
4. Percentage total body fat mass by DXA
5. Appetite score using visual analog scale (VAS)
6. Attention bias to highly palatable images
7. Energy intake at buffet meal
8. Free living physical activity by accelerometry
9. Metabolic syndrome markers (waist circumference, systolic and diastolic blood pressure, lipids, fasting plasma glucose level)
10. Fasting plasma insulin and HOMA-IR index
11. 2-hour oral glucose tolerance test (OGTT) insulin and glucose measurements
12. Hemoglobin A1C
13. Plasma GI hormones (GLP-1 and PYY) during OGTT
14. Weight related quality of life (QoL) score
15. Beck Depression Inventory total score
16. Body-Esteem Scale Score for Adolescents and Adults
17. Columbia Suicide Severity Rating Scale
18. Secretome analysis
19. Stool microbiome analysis

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, 12-20.999 years at screening visit
2. 12 months or more status-post vertical sleeve gastrectomy with a maximum of 10 years after surgery
3. BMI 30 kg/m2 or greater than or equal to 95th percentile for age and sex
4. In good general health as evidenced by medical history
5. Ability to take subcutaneous medication and be willing to adhere to the daily subcutaneous liraglutide regimen
6. Ability to provide consent/assent before any trial-related activities as required per protocol
7. Stated availability for the duration of the study

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current or recent (within 3 months of start of study drug initiation) use of weight loss medications such as phentermine, topiramate, lisdexamfetamine (prescribed specifically for weight loss; when prescribed for ADHD and dose is stable for last 3 months this medication will be allowed), orlistat, and naltrexone HCl/bupropion HCl, or liraglutide
2. Weight of more than 450 lbs. (because Dual-Energy X-ray Absorptiometry (DXA) scanning cannot be done in those exceeding this weight)
3. Current use of insulin or sulfonylurea or other medication affecting insulin secretion or GLP1 clearance such as a DPPIV inhibitor
4. Weight loss of more than 3% of body weight in the past 2 months
5. Current pregnancy, desire to become pregnant within study period, current lactation or, if sexually active, not willing to use adequate contraceptive measures
6. History of recurrent pancreatitis (greater than 2 episodes)
7. History of chronic kidney disease (eGFR <60)
8. History of gastroparesis
9. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
10. History of prior metabolic and bariatric surgery other than vertical sleeve gastrectomy
11. Current or prior use of any GLP-1 agonist medication during the 6 months before screening, including liraglutide.
12. Known or suspected allergy to trial medication, excipients, or related products
13. Treatment with another investigational drug or other experimental intervention within 3 months prior to enrollment in this trial
14. Individuals who have current substance abuse or a DSM 5 Axis I psychiatric disorder or DSM Axis II Mental Retardation diagnosis that in the opinion of the investigators would impede competence, compliance, or participation in the study
15. Suicidal ideation type 4 or 5, history of past suicide attempt, and suicidal behavior in the past month
16. Presence of a major medical illness not listed above

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data for all IPD that underlie results in a publication will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting 6 months after publication or after 1 year following study closure.
Access Criteria: Data will be stored in NIH CTDB and will be made available to university-based researchers on reasonable request to the Principal Investigator following establishment of a data sharing agreement. Afterwards, the data will be deidentified and transferred to DASH

REFERENCES:
- [Background] Kelly AS, Auerbach P, Barrientos-Perez M, Gies I, Hale PM, Marcus C, Mastrandrea LD, Prabhu N, Arslanian S; NN8022-4180 Trial Investigators. A Randomized, Controlled Trial of Liraglutide for Adolescents with Obesity. N Engl J Med. 2020 May 28;382(22):2117-2128. doi: 10.1056/NEJMoa1916038. Epub 2020 Mar 31. PMID 32233338
- [Background] Pi-Sunyer X, Astrup A, Fujioka K, Greenway F, Halpern A, Krempf M, Lau DC, le Roux CW, Violante Ortiz R, Jensen CB, Wilding JP; SCALE Obesity and Prediabetes NN8022-1839 Study Group. A Randomized, Controlled Trial of 3.0 mg of Liraglutide in Weight Management. N Engl J Med. 2015 Jul 2;373(1):11-22. doi: 10.1056/NEJMoa1411892. PMID 26132939
- [Background] Inge TH, Courcoulas AP, Jenkins TM, Michalsky MP, Helmrath MA, Brandt ML, Harmon CM, Zeller MH, Chen MK, Xanthakos SA, Horlick M, Buncher CR; Teen-LABS Consortium. Weight Loss and Health Status 3 Years after Bariatric Surgery in Adolescents. N Engl J Med. 2016 Jan 14;374(2):113-23. doi: 10.1056/NEJMoa1506699. Epub 2015 Nov 6. PMID 26544725
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000241-CH.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 43 participants were screened in person. A total of 34 participants were found eligible and prescribed liraglutide
Groups:
- Liraglutide: Treated with Liraglutide
  Liraglutide: Liraglutide by subcutaneous injection administered daily. Dose was initiated at 0.6mg per day and increased to a maximum of 3.0 mg per day as tolerated.
Period: Overall Study
Arm/Group | Liraglutide
Started | 34
Completed | 31
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Liraglutide
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.97 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 7
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 34
Suboptimal response to sleeve gastrectomy (<20% BMI rediction at BMI nadir [Count of Participants; unit: Participants] | 8
BMI [Mean (Standard Deviation); unit: kg/m2] — Body mass index calculated as the weight in kg divided by the height in meters squared (kg/m2)
  kg/m2 | 41.2 (7.7)
Body Mass Index Z-score [Mean (Standard Deviation); unit: Z-score] — Body Mass Index (BMI) standard deviation score for age and sex, calculated according to the US Centers for Disease Control standards. The BMI (weight in kg divided by the square of height in cm) is converted to a Z-score where a value of 0 represents the population mean for a give age and sex assigned at birth (male or female). Values are considered normal when BMI Z-score is between -1 and 1. Obesity is defined as BMI Z-score >1.64. Reductions in BMI Z-scores are good outcomes for people with obesity.
  Reference: Kuczmarski et a;. Vital Health Stat 11. 2002:1-190.
  Z-score | 2.70 (0.95)
Weight [Mean (Standard Deviation); unit: kg] | 114.9 (21.0)
Years after vertical sleeve gastrectomy was performed [Mean (Standard Deviation); unit: years] | 2.12 (1.13)

OUTCOME MEASURES:

1. Primary Outcome: Cohen's d (the Standardized Mean Difference)
Description: The change in BMI (kg/m2) measured from the baseline visit to the week 16 visit was used to inform a power calculation for a subsequent randomized controlled trial, assuming no change in BMI for the placebo group and the change in BMI that was found in this study at 16 weeks for the liraglutide group. There is no statistical analysis associated with this result.
Time Frame: 16 weeks
Population: Intent to treat sample
Measure: Number (95% Confidence Interval); unit: cohen's d
Arm/Group | Liraglutide
Number analyzed (Participants) | 34
cohen's d | 2.145 [1.72 to 2.55]

2. Secondary Outcome: Change in Fat Mass
Description: Change in fat mass (in kg) from baseline to the week 16 visit using the full intention to treat sample with last observation carried forward if data were missing
Time Frame: 16 weeks
Population: Intent to treat analysis using last observation carried forward. Note one participant did not have data at baseline.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide
Number analyzed (Participants) | 33
kg | -3.2 (3.4)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Superiority; p < 0.001, t-test, 2 sided; Paired t-test, 32 degrees of freedom (one participant did not have baseline DEXA data so could not be included; Mean Difference (Final Values) = -3.2, Standard Deviation 3.4

3. Secondary Outcome: Change in BMI
Description: The change in BMI (kg/m2) from baseline to the week 16 visit using the full intention to treat sample with last observation carried forward if data were missing
Time Frame: 16 weeks
Population: Intent to treat analysis using last observation carried forward
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Liraglutide
Number analyzed (Participants) | 34
kg/m2 | -1.7 (1.5)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Superiority; p < 0.001, t-test, 2 sided; Paired t-test, 33 degrees of freedom; Mean Difference (Final Values) = -1.7, Standard Deviation 1.5

4. Secondary Outcome: Change in Body Mass Index Z-score
Description: The change in Body Mass Index Z-score (standard deviation score for age and sex based on US Centers for Disease Control Standards from baseline to the week 16 visit using the full intention to treat sample with last observation carried forward if data were missing. Please see description for Body Mass Index Z-score in baseline information section for more details on calculation of Body Mass Index Z-score.
Time Frame: 16 weeks
Population: Intention to treat sample with last observation carried forward
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Liraglutide
Number analyzed (Participants) | 34
Z-score | -0.2 (0.1)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Superiority; p < 0.001, t-test, 2 sided; Paired t-test, 33 degrees of freedom; Mean Difference (Final Values) = -0.2, Standard Deviation 0.1

5. Secondary Outcome: Change in Body Weight
Description: The change in body weight (kg) from baseline to the week 16 visit using the full intention to treat sample with last observation carried forward if data were missing
Time Frame: 16 weeks
Population: Intent to treat sample with last observation carried forward
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide
Number analyzed (Participants) | 34
kg | -4.4 (4.4)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Superiority — Paired t-test; p < 0.001, t-test, 2 sided; Paired t-test, 33 degrees of freedom; Mean Difference (Final Values) = -4.4, Standard Deviation 4.4

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events were collected using a detailed checklist for commonly observed adverse events with liraglutide treatment, supplemented by reports from clinician interviews.
Arm/Group | Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 19/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=34)
Dyspepsia (Gastrointestinal disorders) | 8 (16)
Constipation (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 4 (8) — Low Energy
Dizziness (General disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT04883346/Prot_SAP_000.pdf
  • Informed Consent Form: Consent that Parents signed (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04883346/ICF_003.pdf
  • Informed Consent Form: Assent that children signed (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT04883346/ICF_004.pdf